CLINICAL TRIAL: NCT05481554
Title: Composition and Function of Gut Microbiota in Porto-sinusoidal Vascular Disease Associated With Variable Common Immunodeficiency
Acronym: MI-MVPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211408; 2021-A02267-34 (Other: ANSM)
Record Dates: First submitted 2022-06-10; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Common Variable Immunodeficiency; Vascular Diseases
Keywords: Common variable immunodeficiency; Porto-sinusoidal vascular disease; Gut microbiota
MeSH Terms: conditions — Common Variable Immunodeficiency; Vascular Diseases; Idiopathic Noncirrhotic Portal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Common variable immunodeficiency with enteropathy: 20 patients with a common variable immunodeficiency associated to enteropathy will be recruited in the study and will be compared with patients with a common variable immunodeficiency associated to enteropathy and porto-sinusoidal vascular disease
  Interventions: Biological: Stool sample
- Common variable immunodeficiency with enteropathy and porto-sinusoidal vascular disease: 20 patients with common variable immunodeficiency associated to enteropathy and porto-sinusoidal vascular disease will be recruited in the study and will be compared with patients with a common variable immunodeficiency associated to enteropathy
  Interventions: Biological: Stool sample

INTERVENTIONS:
Biological: Stool sample — Only 1 stool sample will be collected during the patient hospitalisation scheduled within standard care.

SUMMARY:
This aim of this study is the evaluation of the gut microbiota imbalance occurrence and its characterization in patients with common variable immunodeficiency associated to an enteropathy with or without porto-sinusoidal vascular disease.

DETAILED DESCRIPTION:
Common variable immunodeficiency (CVID) is the most common symptomatic humoral deficiency in adults and is accompanied by digestive symptoms. It is associated with intestinal dysbiosis and half of the patients exert a clinical digestive disease, called enteropathy. Hepatic complications characterized by porto-sinusoidal vascular disease are observed in 10% of the CVID patients. This complication is associated with a high morbi-mortality. In our center experience and in the literature, clinical occurrence of enteropathy and hepatic disease are highly correlated. Considering (i) the anatomical link between the intestinal tractus and the portal circulation, (ii) the clinical correlation between enteropathy and the liver disease and (iii) the established relation between gut microbiota and alcoholic cirrhosis, we speculate that patients whom develop portosinusoidal complications exert a peculiar intestinal dysbiosis.

This study could contribute to a better understanding of the hepatic disease development, hence allowing us to suggest novel therapies based on gut microbiota modification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with a common variable immunodeficiency according to immune deficiencies classification associated with :

  * enteropathy and porto-sinusoidal vascular disease
  * enteropathy without porto-sinuoidal vascular disease
* Subject with health insurance (AME excepted)
* Verbal agreement to participate at the study

Exclusion Criteria:

- Laxatives in the month preceding stool sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with common variable immunodeficiency associated with enteropathy and with or without portosinusoidal vascular disease.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a dysbiosis | Day 7
  Evaluate the occurrence of dysbiosis and characterize gut microbiota (function and composition) by genomic (16S) and metabolomic (short chain fatty acids, bile acids, tryptophan metabolites) analyses from stool samples of patients with a common variable immunodeficiency with only enteropathy compared to patients with common variable immunodeficiency with enteropathy and porto-sinusoidal vascular disease
Characterization of gut microbiota | Day 7
  Evaluate the occurrence of dysbiosis and characterize gut microbiota (function and composition) by genomic (16S) and metabolomic (short chain fatty acids, bile acids, tryptophan metabolites) analyses from stool samples of patients with a common variable immunodeficiency with only enteropathy compared to patients with common variable immunodeficiency with enteropathy and porto-sinusoidal vascular disease

SECONDARY OUTCOMES:
Fecal calprotectin measurement | Day 7
  Evaluate the contribution of fecal calprotectin measurement at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jehane FADLALLAH, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Immunologie Clinique Hôpital Saint Louis, Paris, France